CLINICAL TRIAL: NCT06148194
Title: Efficacy of Physiological Saline and Probiotics (LiveSpo Navax) in Preventing Respiratory Diseases in Children Aged 2-5, in Son Tay Province, Hanoi
Brief Title: Efficacy of Probiotics (LiveSpo Navax) in Preventing Respiratory Diseases in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anabio R&D (Industry)
Collaborators: Hanoi Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: TNLS.2023.NP; No. 202/HDDD-VKC (Other: Hanoi Medical University)
Record Dates: First submitted 2023-11-18; First posted 2023-11-28 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Respiratory Disease; Respiratory Infections in Children
Keywords: Acute respiratory infection; Prevention; Nasal-spraying probiotics; Bacillus spores; Children; Viruses; Bacterial co-infection
MeSH Terms: conditions — Respiration Disorders; Virus Diseases

STUDY DESIGN:
Intervention Model Description: Blind, randomized, and controlled clinical trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: LiveSpo Navax and placebo 0.9% NaCl physiological saline are indistinguishable regarding taste and smell. The color and turbidity of LiveSpo Navax suspension are unrecognizable to investigators, trainers, child caregivers, children's parents, and children due to opaque plastic container. Only the PI and a data analyst are aware of the group codes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Placebo Comparator): The control group receives 0.9% NaCl physiological saline. Caregivers will spray the children twice daily (morning and afternoon), administering 2 sprays in each nostril and 2 sprays in the throat each time (totally 6 sprays each time) for a continuous period of 4 weeks, starting from the time of study participation.
  Interventions: Drug: 0.9% NaCl physiological saline
- Probiotic 1 (Experimental): The Probiotic 1 group receives LiveSpo® Navax product which is NaCl 0.9% plus B. subtilis and B. clausii at 1 billion CFU/mL x 30 mL. Caregivers will spray the children twice daily (morning and afternoon), administering 2 sprays in each nostril and 2 sprays in the throat each time (totally 6 sprays each time) for a continuous period of 4 weeks, starting from the time of study participation.
  Interventions: Combination Product: Probiotic 1
- Probiotic 2 (Experimental): The Probiotic 2 group receives LiveSpo® Navax Kid product which is NaCl 0.9% plus B. subtilis and B. clausii at 0.6 billion CFU/mL x 30 mL. Caregivers will spray the children twice daily (morning and afternoon), administering 2 sprays in the nose and 2 sprays in each nostril, and 2 sprays in the throat each time (totally 6 sprays each time) for a continuous period of 4 weeks, starting from the time of study participation.
  Interventions: Combination Product: Probiotic 2

INTERVENTIONS:
Drug: 0.9% NaCl physiological saline — Nasal-spraying 0.9% NaCl physiological saline is prepared by extracting 5 mL from 0.9% NaCl intravenous infusion 500 mL PP bottle (B.Braun, Germany, product declaration No. Nasal-spraying 0.9% NaCl physiological saline is prepared by extracting 30 mL from 0.9% NaCl intravenous infusion 500 mL PP bottle (B.Braun, Germany, product declaration No. VD-32732-19), and then pouring it into the same opaque plastic spraying 30 mL-bottle that is used for probiotic 1 and 2.
  Other Names: Registration number: VD-32723-19
  Arms: Control
Combination Product: Probiotic 1 — In Vietnam, LiveSpo Navax is manufactured as a Class-A medical device (Product declaration: No. 210001337/PCBA-HN) in accordance with manufacturing standards approved by the Hanoi Health Department, Ministry of Health, Vietnam (Certificate No. YT117-19), and ISO 13485:2016. LiveSpo Navax product is prepared in the form of NaCl 0.9% plus B. subtilis and B. clausii at 1 billion CFU/mL x 30 mL.
  Other Names: Registration number: No.210001337/PCBA-HN
  Arms: Probiotic 1
Combination Product: Probiotic 2 — In Vietnam, LiveSpo Navax Kid is manufactured as a Class-A medical device (Product declaration: No. 220002534/PCBA-HN) in accordance with manufacturing standards approved by the Hanoi Health Department, Ministry of Health, Vietnam (Certificate No. YT117-19), and ISO 13485:2016. LiveSpo Navax Kid is prepared in the form of NaCl 0.9% plus B. subtilis and B. clausii at 0.6 billion CFU/mL x 30 mL.
  Other Names: Registration number: No. 220002534/PCBA-HN
  Arms: Probiotic 2

SUMMARY:
Acute respiratory infections are common diseases worldwide with the highest incidence and mortality rates, especially among children. Currently, the prevention of acute respiratory infections in children still faces certain limitations. Although there is a vaccine available for influenza, there are no vaccines yet for RSV and adenovirus in children, and influenza vaccination needs to be repeated annually to achieve optimal effectiveness. Therefore, maintaining respiratory and throat hygiene is essential for both treatment and prevention, ensuring respiratory health for children and reducing the risk of bacterial co-infections. In recent years, preventive strategies for respiratory inflammation have garnered increasing attention, with probiotics being shown to have the potential to support treatment and prevention & reduce the risk of recurrent respiratory infections, thus decreasing reliance on antibiotics. Here, the investigators propose that direct nasal spraying of probiotics may be safe and effective in preventing respiratory diseases.

The aim of the study is to evaluate the effectiveness of two types of nasal- praying Bacillus probiotics including LiveSpo Navax (1 billion/mL x 30 mL B. subtilis and B. clausii) and LiveSpo Navax Kid (0.6 billion/mL x 30 mL B. subtilis and B. clausii) in preventing respiratory diseases. Study Population: The sample size is 600. Description of Sites: The study is conducted at preschools in Son Tay Province, Hanoi, Vietnam.

Description of Study Intervention: A total of 600 eligible children are randomly divided into three groups (n = 200/group each). Children in the Control group received 0.9% NaCl physiological saline twice daily (morning and afternoon), with 2 sprays in each nostril and 2 sprays in the throat each time (totally 6 sprays each time), continuously for four weeks. Children in the Probiotic 1 group receive LiveSpo Navax product, and children in the Probiotic 2 group receive LiveSpo Navax Kid, with the same dosage and frequency as the Control group.

Study Duration: 12 months.

DETAILED DESCRIPTION:
Acute respiratory infections are common diseases worldwide with the highest incidence and mortality rates, especially among children. Vietnam is one of the 15 countries with the highest pneumonia rates in the world, with an estimated 2.9 million cases occurring annually. The age group most susceptible to acute respiratory infections is children under 5 years old, especially bronchiolitis, which often occurs in children under 2 years old. The incidence of acute respiratory infections varies with the seasons, with the highest prevalence of viral respiratory infections typically occurring during the winter and spring. In tropical regions, acute respiratory infections are more common during the rainy months, while in temperate regions, they are more prevalent during the winter months. Approximately 30-60% of outpatient visits for medical care are due to acute respiratory infections.

Currently, the prevention of acute respiratory infections in children still faces certain limitations. Although there is a vaccine available for influenza, there are no vaccines yet for RSV and adenovirus in children, and influenza vaccination needs to be repeated annually to achieve optimal effectiveness. Therefore, maintaining respiratory and throat hygiene is essential for both treatment and prevention, ensuring respiratory health for children and reducing the risk of bacterial co-infections. Here, the investigators propose that direct nasal spraying of probiotics may be a safe and effective method for preventing respiratory diseases.

The objective of this study is to investigate the safety and preventive effects of two types of nasal-spraying Bacillus probiotics: LiveSpo Navax (1 billion/mL x 30 mL B. subtilis and B. clausii) and LiveSpo Navax Kid (containing 0.6 billion/mL x 30 mL B. subtilis and B. clausii) in preventing respiratory diseases in healthy children attending preschools. The investigators will evaluate the preventive efficacy in terms of reducing the number of respiratory disease episodes and the number of courses of antibiotics in children after 2 weeks and 4 weeks of using LiveSpo Navax and LiveSpo Navax Kid.

A randomized, double-blind, and controlled clinical trial will be conducted. Parents of the will be required to provide various information about their children, including their full names, sex, ages, respiratory infection history, and history of antibiotic use... After obtaining informed consent, 600 children will be randomly assigned to three groups (n = 200/group): the control group (referred to as the "Control" group) will receive 0.9% NaCl physiological saline, the experimental group 1 (referred to as the "Probiotic 1" group) will receive the probiotic LiveSpo Navax product, and the experimental group 2 (referred to as the "Probiotic 2" group) will receive the probiotic LiveSpo Navax Kid. Children will be provided with coded nasal sprays in blinded samples to ensure the objectivity of the study. Clinical examinations and monitoring will be conducted after 2 weeks and 4 weeks of the experiment. Nasopharyngeal samples will be collected at the same time as the clinical examinations to assess the presence of probiotic spores in the children's nasal mucosa. During the trial, children's typical clinical symptoms of respiratory tract infections are monitored, including runny nose, stuffy nose, sneezing, sore throat, cough, and fatigue. Data is collected on the number of cold or illness episodes, the average duration of each illness episode, the number of days absent from school, and medication history after 2 weeks and 4 weeks of participating in the study. The children's health conditions are observed by caregivers, and the information is recorded in medical records. During this study, parents or caregivers are asked to refrain from giving their children other probiotics, whether via nasal spray or oral administration, and to avoid cleaning their children's noses with other 0.9% NaCl physiological saline sprayers. Data collection and statistical analysis will involve collecting individual medical records and systematically organizing the children's information into a dataset.

The prevention efficacy of LiveSpo Navax product (Probiotic 1 group) and LiveSpo Navax Kid (Probiotic 2 group) is evaluated and compared to 0.9% NaCl physiological saline (Control group) based on the following clinical and survey criteria: (i) reduction in the percentage (%) of children with respiratory infections; (ii) reduction in the number of colds, illnesses, or respiratory tract infections in children; (iii) reduction in the duration of medication usage and the number of medication episodes in the treatment of respiratory diseases. Tabular analysis is performed on dichotomous variables using the χ2 test or Fisher's exact test when the expected value of any cell is below five. Continuous variables are compared using either the t-test or the Mann-Whitney test when the data is not normally distributed. Statistical and graphical analyses are conducted using GraphPad Prism v8.4.3 software (GraphPad Software, CA, USA). The significance level for all analyses is set at p < 0.05.

Detection of B. subtilis ANA4 and B. clausii ANA39 in nasopharyngeal samples was conducted at 2 weeks and 4 weeks using real-time PCR with SYBR Green following the ISO 17025:2017 guidelines. This testing was performed at the Spobiotic Research Center.

ELIGIBILITY:
Inclusion Criteria:

* Children (male/female) aged from 2 to 5 years, currently attending a preschool.
* Parents of the pediatric agree to participate in the study, explain, and sign the research consent form.

Exclusion Criteria:

* Children with a history of nasal reconstructive surgery, nasal ulcers, or nasal polyps.
* Children with a history of congenital immunodeficiency or infectious diseases (e.g., HIV).
* Children who regularly use products that may affect the research outcomes (e.g., immunosuppressive/immunostimulant drugs, pain relievers/anti-inflammatory drugs, anti-cough/expectorant drugs, antihistamines, or other probiotics) within 4 weeks before the start of the study.
* Children with co-morbidities that affect cognition and perception.

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 600 (Actual)
Dates: Start 2024-01-02 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-10-23 (Actual)

PRIMARY OUTCOMES:
Percentage of children with respiratory infections | Days 0, 14, and 28
  Percentage (%) of children with respiratory infections (runny nose, tonsillitis, rhinosinusitis, hoarseness, stuffy nose, sneezing, sore throat, cough, feeling tired...) after 2 weeks and 4 weeks of participating in the study
Incidence of medication intakes (%) | Weeks 1-2 and 3-4
  Incidence of medication intakes (%) including antibiotics, cough suppressants/expectorants, anti-inflammatory drugs, antihistamines, antipyretics... between weeks 1-2 and weeks 3-4.

SECONDARY OUTCOMES:
The number of episodes of children with cold/illness/respiratory tract infections. | 2 weeks and 4 weeks
  The number of episodes of children with cold/illness/respiratory tract infections after 2 weeks and after 4 weeks of participating in the study
Duration of illness | 2 weeks and 4 weeks
  The average number of days per episode of cold/illness/respiratory tract infections at 2 weeks and after 4 weeks of participating in the study
Duration of school absence | 2 weeks and 4 weeks
  The average number of days children have to be absent from school due to cold/illness/respiratory tract infections at 2 weeks and after 4 weeks of participating in the study
Duration of respiratory tract disease treatment | 2 weeks and 4 weeks
  The average number of days children undergo treatment for each respiratory tract disease (bronchiolitis, pneumonia, pharyngitis, otitis media, asthma...) after 2 weeks and after 4 weeks of participating in the study
Duration of treatment for respiratory tract diseases with each type of medication | 2 weeks and 4 weeks
  The average number of days children undergo treatment with each type of medication (antibiotics, anti-inflammatory, antipyretics, expectorants, infusion, bronchodilators...) after 2 weeks and after 4 weeks of participating in the study
Percentage (%) of children infected with viral and bacterial infections | Days 0, 14, and 28
  Percentage (%) of children infected with viruses (RSV, Flu, Rhinovirus) at days 0, 14, and 28.
  Percentage (%) of children infected with bacteria (M. catarrhalis, H. influenzae, S. pneumoniae) at days 0, 14, and 28.
  Percentage (%) of children infected with viral and bacterial co-infections at days 0, 14, and 28.

OTHER OUTCOMES:
Changes in the nasal microbiome in children at day 28 compared to day 0. | Days 0 and 28
  Changes in alpha, beta diversity, and taxonomy (phylum, family, genus) of nasopharyngeal samples at day 28 compared to day 0.
Changes in pro/anti-inflammatory cytokine levels in nasopharyngeal samples at days 0, 14, and 28 | Day 0, 14, and 28
  Changes in pro/anti-inflammatory cytokine levels (e.g. IL-6, IL-8, IL-10, TNF-alpha...) in nasopharyngeal samples at days 0, 14, and 28

CONTACTS AND LOCATIONS:
Overall Officials: Thu TH Nguyen, Assoc. Prof., Principal Investigator — Hanoi Medical University; Anh TV Nguyen, Assoc. Prof., Principal Investigator — Spobio Research Center, Anabio R&D
Locations (1):
- Son Tay Province, Hanoi, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Data or samples share that will be coded, with no PHI include. Approval of the request and execution of all applicable agreements (i.e. a material transfer agreement) are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research and will be provided following review and approval of a study protocol, informed consent form (ICF), and clinical study reports (CSR). For more information or to submit a request, please contact anabio.rd2021@gmail.com

REFERENCES:
- [Background] Michelow IC, Olsen K, Lozano J, Rollins NK, Duffy LB, Ziegler T, Kauppila J, Leinonen M, McCracken GH Jr. Epidemiology and clinical characteristics of community-acquired pneumonia in hospitalized children. Pediatrics. 2004 Apr;113(4):701-7. doi: 10.1542/peds.113.4.701. PMID 15060215
- [Background] Shahbazi R, Yasavoli-Sharahi H, Alsadi N, Ismail N, Matar C. Probiotics in Treatment of Viral Respiratory Infections and Neuroinflammatory Disorders. Molecules. 2020 Oct 22;25(21):4891. doi: 10.3390/molecules25214891. PMID 33105830
- [Background] Greenwood B. The epidemiology of pneumococcal infection in children in the developing world. Philos Trans R Soc Lond B Biol Sci. 1999 Apr 29;354(1384):777-85. doi: 10.1098/rstb.1999.0430. PMID 10365403
- [Background] Shi T, McAllister DA, O'Brien KL, Simoes EAF, Madhi SA, Gessner BD, Polack FP, Balsells E, Acacio S, Aguayo C, Alassani I, Ali A, Antonio M, Awasthi S, Awori JO, Azziz-Baumgartner E, Baggett HC, Baillie VL, Balmaseda A, Barahona A, Basnet S, Bassat Q, Basualdo W, Bigogo G, Bont L, Breiman RF, Brooks WA, Broor S, Bruce N, Bruden D, Buchy P, Campbell S, Carosone-Link P, Chadha M, Chipeta J, Chou M, Clara W, Cohen C, de Cuellar E, Dang DA, Dash-Yandag B, Deloria-Knoll M, Dherani M, Eap T, Ebruke BE, Echavarria M, de Freitas Lazaro Emediato CC, Fasce RA, Feikin DR, Feng L, Gentile A, Gordon A, Goswami D, Goyet S, Groome M, Halasa N, Hirve S, Homaira N, Howie SRC, Jara J, Jroundi I, Kartasasmita CB, Khuri-Bulos N, Kotloff KL, Krishnan A, Libster R, Lopez O, Lucero MG, Lucion F, Lupisan SP, Marcone DN, McCracken JP, Mejia M, Moisi JC, Montgomery JM, Moore DP, Moraleda C, Moyes J, Munywoki P, Mutyara K, Nicol MP, Nokes DJ, Nymadawa P, da Costa Oliveira MT, Oshitani H, Pandey N, Paranhos-Baccala G, Phillips LN, Picot VS, Rahman M, Rakoto-Andrianarivelo M, Rasmussen ZA, Rath BA, Robinson A, Romero C, Russomando G, Salimi V, Sawatwong P, Scheltema N, Schweiger B, Scott JAG, Seidenberg P, Shen K, Singleton R, Sotomayor V, Strand TA, Sutanto A, Sylla M, Tapia MD, Thamthitiwat S, Thomas ED, Tokarz R, Turner C, Venter M, Waicharoen S, Wang J, Watthanaworawit W, Yoshida LM, Yu H, Zar HJ, Campbell H, Nair H; RSV Global Epidemiology Network. Global, regional, and national disease burden estimates of acute lower respiratory infections due to respiratory syncytial virus in young children in 2015: a systematic review and modelling study. Lancet. 2017 Sep 2;390(10098):946-958. doi: 10.1016/S0140-6736(17)30938-8. Epub 2017 Jul 7. PMID 28689664
- [Background] Domachowske JB, Anderson EJ, Goldstein M. The Future of Respiratory Syncytial Virus Disease Prevention and Treatment. Infect Dis Ther. 2021 Mar;10(Suppl 1):47-60. doi: 10.1007/s40121-020-00383-6. Epub 2021 Mar 3. PMID 33656652
- [Background] Tiurin EA. [Effect of the use of dysentery divaccine as therapy in experimental radiation sickness on the immune response to heterologous antigens]. Radiobiologiia. 1982 May-Jun;22(3):395-8. No abstract available. Russian. PMID 7122849
- [Background] Lee NK, Kim WS, Paik HD. Bacillus strains as human probiotics: characterization, safety, microbiome, and probiotic carrier. Food Sci Biotechnol. 2019 Oct 8;28(5):1297-1305. doi: 10.1007/s10068-019-00691-9. eCollection 2019 Oct. PMID 31695928
- [Background] Tran DM, Tran TT, Phung TTB, Bui HT, Nguyen PTT, Vu TT, Ngo NTP, Nguyen MT, Nguyen AH, Nguyen ATV. Nasal-spraying Bacillus spores as an effective symptomatic treatment for children with acute respiratory syncytial virus infection. Sci Rep. 2022 Jul 20;12(1):12402. doi: 10.1038/s41598-022-16136-z. PMID 35858943
- [Background] Tran TT, Phung TTB, Tran DM, Bui HT, Nguyen PTT, Vu TT, Ngo NTP, Nguyen MT, Nguyen AH, Nguyen ATV. Efficient symptomatic treatment and viral load reduction for children with influenza virus infection by nasal-spraying Bacillus spore probiotics. Sci Rep. 2023 Sep 8;13(1):14789. doi: 10.1038/s41598-023-41763-5. PMID 37684332